CLINICAL TRIAL: NCT03535948
Title: Outcome of Hodgkin Lymphoma Patients Over Than 60 Years Treated by Chemotherapy and/or Radiotherapy: a Retrospective Study
Brief Title: Elderly Hodgkin Lymphoma Patients Treated With Chemoradiotherapy
Acronym: HODGSA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS2016/hodgSA-CLEMENT-F/AS
Record Dates: First submitted 2018-04-24; First posted 2018-05-24 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-05

CONDITIONS: Hodgkin Lymphoma, Adult
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Outcome of Hodgkin lymphoma patients over than 60 years treated by chemotherapy and/or radiotherapy: retrospective analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients over than 60 years
* Newly diagnosed Hodgkin lymphoma

Exclusion Criteria:

* Data not available

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Hodgkin lymphoma patients over 60 years treated between 2000 and 2013 by chemotherapy and/or radiotherapy in two university hospitals in France
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Time between diagnosis and progression or death - up to 100 weeks
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months

CONTACTS AND LOCATIONS:
Overall Officials: Lauriane Filliatre-Clement, Principal Investigator — CHRU Nancy
Locations (2):
- France (2):
  - CHU Dijon, Dijon
  - CHRU Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No